CLINICAL TRIAL: NCT06178055
Title: A Phase 2, Double-masked, Randomized, Sham-controlled, Multiple-dose Study of the Efficacy and Safety of Intravitreal KUS121 in the Treatment of Non-Arteritic Central Retinal Artery Occlusion (CRAO)
Brief Title: A Study of the Efficacy and Safety of KUS121 in Participants With Acute Non-Arteritic Central Retinal Artery Occlusion (CRAO)
Acronym: GION
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kyoto Drug Discovery and Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KDK-1101-02
Record Dates: First submitted 2023-12-01; First posted 2023-12-20 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Central Retinal Artery Occlusion
MeSH Terms: conditions — Retinal Artery Occlusion | interventions — KUS121

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- KUS121 high dose group (Experimental)
  Interventions: Drug: KUS121 high dose
- KUS121 low dose group (Experimental)
  Interventions: Drug: KUS121 low dose
- Control group (Sham Comparator)
  Interventions: Drug: Sham procedure

INTERVENTIONS:
Drug: KUS121 high dose — Participants will receive KUS121 high dose intravitreal (IVT) injection once on each of 3 consecutive days (Day 1 through Day 3).
  Arms: KUS121 high dose group
Drug: KUS121 low dose — Participants will receive KUS121 low dose intravitreal (IVT) injection once on each of 3 consecutive days (Day 1 through Day 3).
  Arms: KUS121 low dose group
Drug: Sham procedure — Participants will receive a sham procedure that mimics an intravitreal (IVT) injection once on each of 3 consecutive days (Day 1 through Day 3).
  Arms: Control group

SUMMARY:
Central retinal artery occlusion (CRAO) is an ophthalmologic emergency which leads to severe and permanent vision loss. There is no evidence-based therapy for CRAO. The objective of this GION study is to evaluate the efficacy and safety of KUS121 intravitreal (IVT) injection in participants with acute non-arteritic CRAO.

DETAILED DESCRIPTION:
This is a Phase II, double-masked, sham-controlled, multi-center, parallel-group study to evaluate the efficacy and safety of KUS121 intravitreal (IVT) injection in patients with non-arteritic Central Retinal Artery Occlusion (CRAO) diagnosed and treated within 3-48 hours of disease onset. Participants will be randomized to high dose KUS121, low dose KUS121, or sham in a 1:1:1 ratio. Participants will receive daily intravitreal injections of KUS 121 or sham, which mimics an injection, from Day 1 through Day 3. Primary efficacy endpoint is the proportion of participants who gain 15 letters or more in BCVA compared with baseline and will be assessed at Week 12. Safety evaluation will continue until a 12-month follow up.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are willing and able to comply with clinic visits and study-related procedures and able to provide signed informed consent in person or from their legally authorized representative
* Males and females ≥ 20 years of age at that time of providing signed informed consent
* Diagnosed as non-arteritic Central Retinal Artery Occlusion from 3 hours until no more than 48 hours after the onset of significant visual acuity changes
* Best Corrected Visual Acuity (BCVA) Early Treatment Diabetic Retinopathy Study (ETDRS) letter score of 0 to 35 in the study eye at screening prior to enrollment (eyes with 'no light perception' or 'light perception' are to be excluded)
* Retinal thickening or hyper-reflectivity in retinal inner layers in spectral domain optical coherence tomography (SD-OCT), or white turbid edema in fundus examination

Exclusion Criteria:

* Presence of the following conditions in the study eye:

  1. Infection in or around the eye
  2. Uncontrolled intraocular pressure
  3. Abnormality in macula other than CRAO findings
  4. History of macular photocoagulation
  5. Opacity in visual axis preventing fundus examination or fundus imaging (e.g., corneal dystrophy)
  6. Neovascularization of iris and retina
  7. Any inflammatory disease involving the eye
  8. Optic atrophy
  9. Glaucomatous cupping greater than 0.9
  10. Prior vitrectomy
  11. Aphakia with the absence of posterior capsule
  12. Any IVT injection or sub-Tenon's injection within 1 month of screening
  13. Any intraocular surgery or ocular implant within 3 months of screening
  14. Any history of ocular trauma within 3 months of screening
* Thrombolytic, fibrinolytic or prostaglandin E1 systemic treatment within 1 month of screening
* A positive urine pregnancy test on Day 1 prior to study enrollment
* History of allergy or hypersensitivity to KUS121 or a compound with a condensed polycyclic aromatic hydrocarbon skeleton represented by naphthalene and any of excipients of KUS121 product, fluorescein, or any study treatment-related mandatory ingredients that is not amenable to treatment
* Known hypersensitivity to a study treatment procedure, dilating drops, or any of the anesthetic and antimicrobial preparations used by a participant during the study
* Presence of other medical disease, physical or ocular examination finding, or clinical laboratory finding that in the opinion of the Investigator contraindicates the use of an investigational product, might interfere with the evaluation of the efficacy or safety of the study drug, may put the participant at significant risk or might interfere with the participant's ability to participate in the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-04-16 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of study eyes which achieve a gain of 15 ETDRS letters or more in BCVA at Week 12 compared to baseline | At baseline, Week 12
  BCVA: Best-Corrected Visual Acuity; ETDRS: Early Treatment Diabetic Retinopathy Study. A higher ETDRS letter score means a better outcome (better visual acuity).

SECONDARY OUTCOMES:
Proportion of study eyes which achieve a gain of 15 ETDRS letters or more in BCVA at Week 4 compared to baseline | At baseline, Week 4
Proportion of study eyes which achieve a gain of 0.3 Logarithm of Minimum Angle of Resolution (Log MAR) in BCVA at Week 12 compared to baseline | At baseline, Week 12
  BCVA will be recorded using a Logarithm of the Minimum Angle of Resolution (LogMAR) scoring chart. A lower LogMAR score means a better outcome (better visual acuity).
Proportion of study eyes which achieve a gain of 10 ETDRS letters or more in BCVA at Week 12 compared to baseline | At baseline, Week 12
Mean change in BCVA (readable letters and Log MAR) at Week 12 compared to baseline | At baseline, Week 12
Change in retinal thickness from baseline at Week 12 as measured by SD-OCT | At baseline, Week 12
Change in the area of visual field from baseline to Week 12 as measured by Humphrey Field Analyzer | At baseline, Week 12
  The Humphrey Visual Field Analyser test assesses the retina's ability to detect a light stimulus at specific points within the visual field. A higher score means a better outcome (better visual field).
Incidence and Severity of Ocular and Systemic (Non-Ocular) Adverse Events (AEs) | From baseline through Week 48
Patients Reported Outcome | Up to Week 12
  The results of National Eye Institute Visual Function Questionnaire (NEI-VFQ 25) for each group at before, afterwards the disease onset and Week 12. A higher score means a better functioning (better patient-reported visual function).

CONTACTS AND LOCATIONS:
Overall Officials: Kunihiro Musashi, MD., Ph.D., Study Chair — Kyoto Drug Discovery ＆ Development Co., Ltd.
Locations (11):
- United States (11):
  - The Retina Partners, Encino, California
  - Salehi Retina Institute, Inc, Huntington Beach, California
  - Kaiser Permanente Oakland Med Ctr., Oakland, California
  - Florida Retina Institute, Jacksonville, Florida
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Kresge Eye Institute/Wayne State University, Detroit, Michigan
  - NYEE Infirmary of Mount Sinai, New York, New York
  - UH Eye Institute, Cleveland, Ohio
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ikeda HO, Muraoka Y, Hata M, Sumi E, Ikeda T, Nakagawa T, Abe H, Tada H, Morita S, Kakizuka A, Yoshimura N, Tsujikawa A. Safety and effectiveness of a novel neuroprotectant, KUS121, in patients with non-arteritic central retinal artery occlusion: An open-label, non-randomized, first-in-humans, phase 1/2 trial. PLoS One. 2020 Feb 13;15(2):e0229068. doi: 10.1371/journal.pone.0229068. eCollection 2020. PMID 32053676